CLINICAL TRIAL: NCT01707290
Title: A Phase 3, Two-Arm, Rollover Study to Evaluate the Safety of Long Term Ivacaftor Treatment in Subjects 6 Years of Age and Older With Cystic Fibrosis and a Non-G551D CFTR Mutation
Brief Title: Rollover Study of Ivacaftor in Subjects With Cystic Fibrosis and a Non G551D CFTR Mutation
Acronym: KONTINUE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX12-770-112; 2012-000389-39 (EudraCT Number)
Record Dates: First submitted 2012-10-09; First posted 2012-10-16 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ivacaftor (Experimental): Participants who received Ivacaftor 150 milligram (mg) tablet and/or Placebo matched to Ivacaftor tablet orally, every 12 hours (q12h) in the previous study VX11-770-110 (Study 110; NCT01614457), VX12-770-111 (Study 111; NCT01614470) or VX12-770-113 (Study 113; NCT01685801); received Ivacaftor 150 mg tablet q12h in this VX12-770-112 (Study 112; NCT01707290) up to 104 weeks.
  Interventions: Drug: Ivacaftor
- Observational (No Intervention): Participants who received Ivacaftor 150 mg tablet and/or Placebo matched to Ivacaftor tablet, orally, q12h in the previous Study 110 (NCT01614457) or Study 111 (NCT01614470), were observed (did not receive study drug) in this Study 112 (NCT01707290) for up to 2 years.

INTERVENTIONS:
Drug: Ivacaftor — 150 mg tablet, oral use, every 12 hours (q12h)
  Other Names: Kalydeco; VX-770
  Arms: Ivacaftor

SUMMARY:
The purpose of this study is to evaluate the safety of long-term ivacaftor treatment in participants with cystic fibrosis (CF) from Studies 110 (NCT01614457), 111 (NCT01614470), and 113 (NCT01685801).

DETAILED DESCRIPTION:
Ivacaftor is the first Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) modulator to show an improvement in CFTR function and clinical benefit in participants with CF. Results from Phase 3 studies (NCT00909532 [Study 102] and NCT00909727 [Study 103]) showed that ivacaftor is effective in the treatment of participants with CF who have the G551D-CFTR mutation, as evidenced by sustained improvements in CFTR channel function (measured by reduction in sweat chloride concentration) and corresponding substantial, durable improvements in lung function, pulmonary exacerbations, respiratory symptoms, and weight gain. Ivacaftor was also well tolerated, as evidenced by the rates and reasons for premature discontinuation and results of safety assessments.

Ivacaftor (Trade Name Kalydeco; 150 mg tablets) was initially approved in the United States for the treatment of CF in participants 6 years of age and older who have a G551D mutation in the CFTR gene.

ELIGIBILITY:
Inclusion Criteria:

* Participants from Study 110 or Study 111 entering the ivacaftor arm must have completed the assigned study drug treatment duration in the previous study.
* Participants from Study 113 entering the ivacaftor arm must have completed all study related treatments through the Follow-up Visit and met the Study 113 responder criteria during the previous study.
* Participants entering the observational arm must have completed at least 4 weeks of study drug treatment in their previous study (Study 110 or Study 111), must have completed the previous study but do not wish to enroll in the ivacaftor arm, or must have completed the previous study but do not meet the inclusion criteria of the ivacaftor arm.
* Participants of childbearing potential entering the ivacaftor arm must not be pregnant.
* Participants entering the ivacaftor arm must be willing to comply with contraception requirements.

Exclusion Criteria (Ivacaftor Arm Only):

* History of any illness or condition that might confound the results of the study or pose an additional risk in administering ivacaftor to the Participant.
* Use of moderate or strong inhibitors or inducers of cytochrome P450 (CYP) 3A.
* Evidence of cataract or lens opacity at or before the Day 1 Visit.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2013-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Pilewski, MD, Principal Investigator — University of Pittsburgh
Locations (38):
- United States (33):
  - Birmingham, Alabama
  - Palo Alto, California
  - Denver, Colorado
  - Hartford, Connecticut
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Iowa City, Iowa
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - New York, New York
  - Syracuse, New York
  - Valhalla, New York
  - Chapel Hill, North Carolina
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Seattle, Washington
  - Morgantown, West Virginia
  - Madison, Wisconsin
- Leuven, Belgium
- France (2):
  - Montpellier
  - Paris
- United Kingdom (2):
  - Belfast
  - Edinburgh

REFERENCES:
- [Derived] Pilewski JM, De Boeck K, Nick JA, Tian S, DeSouza C, Higgins M, Moss RB. Long-Term Ivacaftor in People Aged 6 Years and Older with Cystic Fibrosis with Ivacaftor-Responsive Mutations. Pulm Ther. 2020 Dec;6(2):303-313. doi: 10.1007/s41030-020-00129-2. Epub 2020 Sep 23. PMID 32965659
- [Derived] Moss RB, Flume PA, Elborn JS, Cooke J, Rowe SM, McColley SA, Rubenstein RC, Higgins M; VX11-770-110 (KONDUCT) Study Group. Efficacy and safety of ivacaftor in patients with cystic fibrosis who have an Arg117His-CFTR mutation: a double-blind, randomised controlled trial. Lancet Respir Med. 2015 Jul;3(7):524-33. doi: 10.1016/S2213-2600(15)00201-5. Epub 2015 Jun 9. PMID 26070913

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 2 arms: Ivacaftor arm and Observational arm. The Ivacaftor arm enrolled subjects from Study VX11-770-110 (NCT01614457), Study VX12-770-111 (NCT01614470) and Study VX12-770-113 (NCT01685801). The Observational arm enrolled subjects from Study VX11-770-110 (NCT01614457) and Study VX12-770-111 (NCT01614470).
Groups:
- Ivacaftor Arm: Participants who received Ivacaftor 150 milligram (mg) tablet and/or Placebo matched to Ivacaftor tablet, every 12 hours (q12h) in the previous study VX11-770-110 (Study 110; NCT01614457), VX12-770-111 (Study 111; NCT01614470) or VX12-770-113 (Study 113; NCT01685801); received Ivacaftor 150 mg tablet orally q12h in this VX12-770-112 (Study 112; NCT01707290) up to 104 weeks.
- Observational Arm: Participants who received Ivacaftor 150 mg tablet and/or Placebo matched to Ivacaftor tablet q12h in the previous Study 110 (NCT01614457) or Study 111 (NCT01614470), were observed (did not receive study drug) in this Study 112 (NCT01707290) for up to 2 years.
Period: Overall Study
Arm/Group | Ivacaftor Arm | Observational Arm
Started | 121 | 4
Completed | 35 | 3
Not Completed | 86 | 1
Not completed — Adverse event (AE) | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal of Consent (Not Due to AE) | 4 | 0
Not completed — Commercial drug available | 60 | 1
Not completed — Other unspecified | 17 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ivacaftor Arm: Participants who received Ivacaftor 150 mg tablet and/or Placebo matched to Ivacaftor tablet, q12h in the previous study VX11-770-110 (Study 110; NCT01614457), VX12-770-111 (Study 111; NCT01614470) or VX12-770-113 (Study 113; NCT01685801); received Ivacaftor 150 mg tablet orally q12h in this VX12-770-112 (Study 112; NCT01707290) up to 104 weeks.
- Total: Total of all reporting groups
Arm/Group | Ivacaftor Arm | Observational Arm | Total
Number analyzed (Participants) | 121 | 4 | 125
Age, Customized [Number; unit: participants]
  6 to 11 years | 21 | 1 | 22
  12 to 17 years | 11 | 1 | 12
  18 years and over | 89 | 2 | 91
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 3 | 64
  Male | 60 | 1 | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) or Serious Adverse Events (SAEs) in Ivacaftor Arm
Description: AE: any untoward medical occurrence in a participants during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or previous condition that has increased in severity or frequency after informed consent form is signed. AE includes serious as well as non-serious AEs. SAE (subset of AE): medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, In-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. TEAEs were defined as adverse events with start date or increased severity on and after the first dose of study drug through Week 108.
Time Frame: Day 1 up to Week 108 (Study 112)
Population: Safety Set included all participants who received at least 1 dose of study drug (Ivacaftor).
Measure: Number; unit: participants
Groups:
- Ivacaftor Arm: Participants who received Ivacaftor 150 mg tablet and/or Placebo matched to Ivacaftor tablet q12h in the previous study VX11-770-110 (Study 110; NCT01614457), VX12-770-111 (Study 111; NCT01614470) or VX12-770-113 (Study 113; NCT01685801); received Ivacaftor 150 mg tablet orally q12h in this VX12-770-112 (Study 112; NCT01707290) up to 104 weeks.
Arm/Group | Ivacaftor Arm
Number analyzed (Participants) | 121
participants
  Participants with TEAEs | 117
  Participants with SAEs | 27

2. Secondary Outcome: Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) at Week 2, 12, 24, 36, 48, 60, 72, 84, 96, and 104
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Hankinson and Wang standards were used to calculate percent predicted FEV1 (for age, gender, and height). The Hankinson standard was used for male participants 18 years and older and female participants 16 years and older. The Wang standard was used for male participants aged 6 to 17 years and for female participants aged 6 to 15 years. Baseline was defined as the most recent measurement before intake of the first dose of study drug (Ivacaftor) in Study 112. Results were planned to be reported for Ivacaftor arm and were stratified by parent study 110, 111 and 113.
Time Frame: Baseline, Week 2, 12, 24, 36, 48, 60, 72, 84, 96 and 104 (Study 112)
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of study drug (Ivacaftor). Here, "Number Analyzed" signifies those participants who were evaluable for this measure at the specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: Percent predicted of FEV1
Groups:
- Ivacaftor Arm: Study 110: Participants who received Ivacaftor 150 mg tablet and/or Placebo matched to Ivacaftor tablet orally, q12h in the previous Study 110; received Ivacaftor 150 mg tablet q12h in this Study 112 up to 104 weeks.
- Ivacaftor Arm: Study 111: Participants who received Ivacaftor 150 mg tablet and/or Placebo matched to Ivacaftor tablet orally, q12h in the previous Study 111; received Ivacaftor 150 mg tablet q12h in this Study 112 up to 104 weeks.
- Ivacaftor Arm: Study 113: Participants who received Ivacaftor 150 mg tablet and/or Placebo matched to Ivacaftor tablet orally, q12h in the previous Study 113; received Ivacaftor 150 mg tablet q12h in this Study 112 up to 104 weeks.
Arm/Group | Ivacaftor Arm: Study 110 | Ivacaftor Arm: Study 111 | Ivacaftor Arm: Study 113
Number analyzed (Participants) | 65 | 35 | 21
Percent predicted of FEV1
  Baseline | 71.8 (20.4) | 78.3 (21.1) | 62.8 (22.2)
  Change at Week 2 | 3.8 (8) | 4.4 (7.7) | 4 (7.2)
  Change at Week 12: number analyzed (Participants) | 63 | 33 | 21
  Change at Week 12 | 5.4 (8.9) | 5.5 (8.3) | 4.9 (6.7)
  Change at Week 24: number analyzed (Participants) | 62 | 34 | 21
  Change at Week 24 | 4.5 (8.4) | 7.1 (8.3) | 4.6 (8.5)
  Change at Week 36: number analyzed (Participants) | 60 | 29 | 20
  Change at Week 36 | 4.4 (7.1) | 7.5 (8.2) | 4.9 (8.2)
  Change at Week 48: number analyzed (Participants) | 58 | 19 | 20
  Change at Week 48 | 4.4 (7.5) | 6.4 (10.7) | 4.9 (9)
  Change at Week 60: number analyzed (Participants) | 58 | 16 | 20
  Change at Week 60 | 4.5 (8.4) | 8.2 (8.3) | 4.5 (8.8)
  Change at Week 72: number analyzed (Participants) | 50 | 13 | 18
  Change at Week 72 | 3.6 (8.9) | 7.8 (9.2) | 5.9 (9.2)
  Change at Week 84: number analyzed (Participants) | 40 | 11 | 16
  Change at Week 84 | 5.4 (13.5) | 7.7 (7.6) | 4.8 (7.2)
  Change at Week 96: number analyzed (Participants) | 28 | 9 | 15
  Change at Week 96 | 4.1 (14.6) | 9.9 (6.4) | 5.9 (8.1)
  Change at Week 104: number analyzed (Participants) | 20 | 9 | 12
  Change at Week 104 | 4.6 (13.2) | 4.9 (5.8) | 6.3 (10)

3. Secondary Outcome: Absolute Change From Baseline in Body Mass Index (BMI) at Week 2,12, 24, 36, 48, 60, 72, 84, 96 and 104
Description: BMI was defined as weight in kg divided by height in m^2. Baseline was defined as the most recent measurement before intake of the first dose of study drug (Ivacaftor) in Study 112. Results were planned to be reported for Ivacaftor arm and were stratified by parent study 110, 111 and 113.
Time Frame: Baseline, Week 2, 12, 24, 36, 48, 60, 72, 84, 96 and 104 (Study 112)
Population: FAS included all participants who received at least 1 dose of study drug (Ivacaftor). Here, "Number analyzed" signifies those participants who were evaluable for this measure at the specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)
Arm/Group | Ivacaftor Arm: Study 110 | Ivacaftor Arm: Study 111 | Ivacaftor Arm: Study 113
Number analyzed (Participants) | 65 | 35 | 21
kilogram per square meter (kg/m^2)
  Baseline | 23.75 (5.63) | 23.15 (5.28) | 24.81 (5.76)
  Change at Week 2 | 0.06 (0.43) | 0.16 (0.47) | 0.07 (0.43)
  Change at Week 12: number analyzed (Participants) | 64 | 35 | 21
  Change at Week 12 | 0.32 (0.59) | 0.39 (0.62) | 0.22 (0.6)
  Change at Week 24: number analyzed (Participants) | 62 | 35 | 21
  Change at Week 24 | 0.43 (0.92) | 0.65 (0.96) | 0.17 (0.91)
  Change at Week 36: number analyzed (Participants) | 60 | 29 | 20
  Change at Week 36 | 0.62 (1.04) | 0.64 (1.07) | 0.02 (1.27)
  Change at Week 48: number analyzed (Participants) | 59 | 19 | 20
  Change at Week 48 | 0.54 (1.39) | 0.58 (1.22) | 0.28 (1.26)
  Change at Week 60: number analyzed (Participants) | 58 | 16 | 20
  Change at Week 60 | 0.72 (1.32) | 0.25 (1.09) | 0.38 (1.22)
  Change at Week 72: number analyzed (Participants) | 51 | 13 | 17
  Change at Week 72 | 1.05 (1.73) | 0.45 (1.34) | 0.22 (1.22)
  Change at Week 84: number analyzed (Participants) | 40 | 11 | 16
  Change at Week 84 | 0.72 (1.51) | 0.33 (1.42) | 0.23 (0.92)
  Change at Week 96: number analyzed (Participants) | 28 | 9 | 16
  Change at Week 96 | 0.49 (1.44) | 0.1 (1.49) | 0.52 (1.28)
  Change at Week 104: number analyzed (Participants) | 20 | 9 | 12
  Change at Week 104 | 0.42 (1.49) | 0.16 (1.37) | 0.88 (1.39)

4. Secondary Outcome: Absolute Change From Baseline in Sweat Chloride at Week 2, 24, 48 and 104
Description: Sweat samples were collected using an approved collection device. Baseline was defined as the most recent measurement before intake of the first dose of study drug (Ivacaftor) in Study 112. Results were planned to be reported for Ivacaftor arm and were stratified by parent study 110, 111 and 113.
Time Frame: Baseline, Week 2, 24, 48 and 104 (Study 112)
Population: FAS included all participants who received at least 1 dose of study drug (Ivacaftor). Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome and "Number Analyzed" signifies those participants who were evaluable for this measure at the specified time point for each arm respectively.
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Ivacaftor Arm: Study 110 | Ivacaftor Arm: Study 111 | Ivacaftor Arm: Study 113
Number analyzed (Participants) | 59 | 33 | 21
millimole per liter (mmol/L)
  Baseline | 60.9 (19.4) | 80.2 (22.8) | 55.7 (22.2)
  Change at Week 2: number analyzed (Participants) | 59 | 31 | 21
  Change at Week 2 | -19.3 (10.7) | -38.4 (27.5) | -4.5 (10.9)
  Change at Week 24: number analyzed (Participants) | 56 | 33 | 20
  Change at Week 24 | -13 (18.4) | -39.2 (27) | 1.1 (15.8)
  Change at Week 48: number analyzed (Participants) | 50 | 19 | 19
  Change at Week 48 | -13.5 (16.2) | -40.6 (26.1) | -1.9 (17.8)
  Change at Week 104: number analyzed (Participants) | 15 | 9 | 11
  Change at Week 104 | -13.7 (22.9) | -32.9 (26.8) | 5.4 (18.1)

5. Secondary Outcome: Absolute Change From Baseline in Respiratory Domain of the Cystic Fibrosis Questionnaire Revised (CFQ-R) at Week 2, 12, 24, 36, 48, 60, 72, 84, 96 and 104
Description: The CFQ-R is a validated participant reported outcome measuring health related quality of life for participants with CF. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), score range: 0-100; higher scores indicating fewer symptoms and better health related quality of life. Baseline was defined as the most recent measurement before intake of the first dose of study drug (ivacaftor) in Study 112. Results were planned to be reported for Ivacaftor arm and were stratified by parent study 110, 111 and 113.
Time Frame: Baseline, Week 2, 12, 24, 36, 48, 60, 72, 84, 96 and 104 (Study 112)
Population: FAS included all participants who received at least 1 dose of study drug (ivacaftor). Here, "Number Analyzed" signifies those participants who were evaluable for this measure at the specified time point for each arm respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ivacaftor Arm: Study 110 | Ivacaftor Arm: Study 111 | Ivacaftor Arm: Study 113
Number analyzed (Participants) | 65 | 35 | 21
units on a scale
  Baseline | 68.6 (21.6) | 72.4 (20.3) | 65.9 (18.8)
  Change at Week 2 | 5.5 (17.9) | 4.5 (17.5) | 13.2 (16.2)
  Change at Week 12: number analyzed (Participants) | 64 | 35 | 21
  Change at Week 12 | 11.6 (18) | 5.7 (18.5) | 13.5 (20)
  Change at Week 24: number analyzed (Participants) | 62 | 35 | 21
  Change at Week 24 | 6.7 (19) | 3.4 (18.7) | 8.5 (14.9)
  Change at Week 36: number analyzed (Participants) | 60 | 29 | 20
  Change at Week 36 | 12.1 (19.3) | 5.7 (13.8) | 7.9 (20.5)
  Change at Week 48: number analyzed (Participants) | 59 | 19 | 20
  Change at Week 48 | 9.5 (17.6) | 4.4 (13.2) | 11.4 (15.7)
  Change at Week 60: number analyzed (Participants) | 57 | 15 | 20
  Change at Week 60 | 7.1 (18.6) | 4.4 (10.9) | 8.6 (19.3)
  Change at Week 72: number analyzed (Participants) | 51 | 13 | 18
  Change at Week 72 | 10.4 (22.2) | 5.6 (11.8) | 8.6 (19)
  Change at Week 84: number analyzed (Participants) | 40 | 11 | 16
  Change at Week 84 | 10.5 (19.5) | 8.8 (14.1) | 4.9 (14.6)
  Change at Week 96: number analyzed (Participants) | 28 | 9 | 16
  Change at Week 96 | 8.8 (21.1) | 0 (9.5) | 9.4 (14.7)
  Change at Week 104: number analyzed (Participants) | 20 | 9 | 12
  Change at Week 104 | 9.2 (14) | 1.9 (8.8) | 19.9 (16)

6. Secondary Outcome: Number of Pulmonary Exacerbations Events
Description: Pulmonary exacerbation events include those events which require treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms. The number of events were reported. Results were planned to be reported for Ivacaftor arm and were stratified by parent study 110, 111 and 113.
Time Frame: Through Week 104 (Study 112)
Population: FAS included all participants who received at least 1 dose of study drug (Ivacaftor).
Measure: Number; unit: pulmonary exacerbation events
Arm/Group | Ivacaftor Arm: Study 110 | Ivacaftor Arm: Study 111 | Ivacaftor Arm: Study 113
Number analyzed (Participants) | 65 | 35 | 21
pulmonary exacerbation events | 47 | 30 | 6

7. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) in Observational Arm
Description: SAE was defined as a medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, In-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event.
Time Frame: up to 2 years (Study 112)
Population: Analysis population included all participants who were included in the observational arm.
Measure: Number; unit: participants
Groups:
- Observational Arm: Participants who received Ivacaftor 150 mg tablet and/or Placebo matched to Ivacaftor tablet, orally, q12h in the previous Study 110 (NCT01614457) or Study 111 (NCT01614470), were observed (did not receive study drug) in this Study 112 (NCT01707290) for up to 2 years.
Arm/Group | Observational Arm
Number analyzed (Participants) | 4
participants | 1

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 108 for Ivacaftor arm; up to 2 years for Observational arm (Study 112)
Description: Non-SAEs were not collected for Observational arm. Only SAEs were planned to be collected for the Observational arm.
Arm/Group | Ivacaftor Arm | Observational Arm
Serious Adverse Events (participants affected / at risk) | 27/121 | 1/4
Other Adverse Events (participants affected / at risk) | 117/121 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ivacaftor Arm (N=121) | Observational Arm (N=4)
Influenza A virus test positive (Investigations) | 1 | 0
Cardiomyopathy acute (Cardiac disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 21 | 1
Gastroenteritis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 0
Pharyngitis bacterial (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ivacaftor Arm (N=121) | Observational Arm (N=0)
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Pallor (Vascular disorders) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seasonal allergy (Immune system disorders) | 4 | 0
Allergy to arthropod bite (Immune system disorders) | 1 | 0
Pyrexia (General disorders) | 17 | 0
Chest pain (General disorders) | 4 | 0
Influenza like illness (General disorders) | 4 | 0
Fatigue (General disorders) | 12 | 0
Chills (General disorders) | 2 | 0
Feeling of body temperature change (General disorders) | 2 | 0
Pain (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 2 | 0
Device leakage (General disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Implant site rash (General disorders) | 1 | 0
Local swelling (General disorders) | 1 | 0
Vaccination site pain (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 0
Anxiety (Psychiatric disorders) | 6 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 3 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Tobacco abuse (Psychiatric disorders) | 1 | 0
Drug dependence (Psychiatric disorders) | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0
Testicular torsion (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 0
Hand fracture (Injury, poisoning and procedural complications) | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 2 | 0
Muscle strain (Injury, poisoning and procedural complications) | 2 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0
Snake bite (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Bacterial test positive (Investigations) | 7 | 0
Forced expiratory volume decreased (Investigations) | 6 | 0
Weight decreased (Investigations) | 5 | 0
C-reactive protein increased (Investigations) | 4 | 0
Haemophilus test positive (Investigations) | 3 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Liver function test abnormal (Investigations) | 3 | 0
Atypical mycobacterium test positive (Investigations) | 2 | 0
Blood pressure increased (Investigations) | 2 | 0
Hepatic enzyme increased (Investigations) | 2 | 0
Body temperature increased (Investigations) | 2 | 0
Pseudomonas test positive (Investigations) | 2 | 0
Vitamin D decreased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Weight increased (Investigations) | 2 | 0
Blood calcium decreased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Crystal urine present (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Flavobacterium test positive (Investigations) | 1 | 0
Influenza A virus test positive (Investigations) | 1 | 0
Streptococcus test positive (Investigations) | 1 | 0
Klebsiella test positive (Investigations) | 1 | 0
Urinary sediment present (Investigations) | 1 | 0
Ultrasound biliary tract abnormal (Investigations) | 1 | 0
Urine analysis abnormal (Investigations) | 1 | 0
Vitamin A decreased (Investigations) | 1 | 0
White blood cells urine positive (Investigations) | 1 | 0
Pulmonary function test decreased (Investigations) | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 41 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 22 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 22 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 17 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 12 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 9 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung hyperinflation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Prolonged expiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 9 | 0
Headache (Nervous system disorders) | 23 | 0
Migraine (Nervous system disorders) | 3 | 0
Dizziness (Nervous system disorders) | 7 | 0
Burning sensation (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0
Hypersomnia (Nervous system disorders) | 1 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0
Blepharospasm (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 2 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 1 | 0
Eye swelling (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Vitreous floaters (Eye disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 3 | 0
Middle ear effusion (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 17 | 0
Constipation (Gastrointestinal disorders) | 17 | 0
Vomiting (Gastrointestinal disorders) | 12 | 0
Abdominal pain (Gastrointestinal disorders) | 12 | 0
Nausea (Gastrointestinal disorders) | 9 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 0
Tooth impacted (Gastrointestinal disorders) | 3 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Dental caries (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0
Toothache (Gastrointestinal disorders) | 2 | 0
Steatorrhoea (Gastrointestinal disorders) | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Defaecation urgency (Gastrointestinal disorders) | 1 | 0
Dental discomfort (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Palatal disorder (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Tooth loss (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Clubbing (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Cushingoid (Endocrine disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 4 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Impaired fasting glucose (Metabolism and nutrition disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Vitamin A deficiency (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 49 | 0
Nasopharyngitis (Infections and infestations) | 21 | 0
Sinusitis (Infections and infestations) | 18 | 0
Viral upper respiratory tract infection (Infections and infestations) | 17 | 0
Gastroenteritis viral (Infections and infestations) | 9 | 0
Upper respiratory tract infection (Infections and infestations) | 15 | 0
Influenza (Infections and infestations) | 7 | 0
Oral candidiasis (Infections and infestations) | 8 | 0
Gastroenteritis (Infections and infestations) | 5 | 0
Acute sinusitis (Infections and infestations) | 4 | 0
Lower respiratory tract infection (Infections and infestations) | 5 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 3 | 0
Bacterial disease carrier (Infections and infestations) | 3 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 3 | 0
Pharyngitis streptococcal (Infections and infestations) | 3 | 0
Rhinitis (Infections and infestations) | 3 | 0
Respiratory tract infection viral (Infections and infestations) | 3 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 3 | 0
Tonsillitis (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 2 | 0
Otitis externa (Infections and infestations) | 2 | 0
Laryngitis (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 2 | 0
Pharyngitis bacterial (Infections and infestations) | 2 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Croup infectious (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Ear lobe infection (Infections and infestations) | 1 | 0
Haemophilus infection (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infected dermal cyst (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Laryngitis viral (Infections and infestations) | 1 | 0
Molluscum contagiosum (Infections and infestations) | 1 | 0
Myringitis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Oesophagitis bacterial (Infections and infestations) | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Vaginitis bacterial (Infections and infestations) | 1 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Nasal abscess (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.